CLINICAL TRIAL: NCT05393778
Title: Accuracy in aChieving Optimum reconstrUction: Measured- vs. Navigation- Techniques in Hip Arthroplasty
Brief Title: Measured vs Navigated Techniques in Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: FormusLab (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3390
Record Dates: First submitted 2021-12-10; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Measured Technique (Experimental): Patients in this group will have pre-operative planning done using the measured technique.
  Interventions: Procedure: Measured Technique
- Navigated Technique (Experimental): Patients in this group will have pre-operative planning done using the navigated technique.
  Interventions: Procedure: Navigated Technique

INTERVENTIONS:
Procedure: Measured Technique — Manual intra-operative checks and tools are used to aid in component placement during surgery.
  Arms: Measured Technique
Procedure: Navigated Technique — IntelliJoint® navigation is an imageless-based navigation system that utilizes a miniature infrared camera and microelectronics to measure hip center of rotation, acetabular inclination and version, leg length, and offset. The device provides accurate real-time data on implant positioning to aid in placement of the components during surgery.
  Arms: Navigated Technique

SUMMARY:
Accurate reconstruction of the native hip parameters following total hip arthroplasty is associated with improved outcome. In order to improve ability for optimum reconstruction, 3-D templating software can be utilized that provide detailed information regarding native anatomy. In order to achieve reconstruction within acceptable parameters as per pre-operative plan, some surgeons propose the use of intra-operative devices that measure component orientation and joint reconstruction ("Measured-THA"), whilst others propose the use of navigation tools ("Navigation-THA). Both techniques have shown superiority compared to the most commonly used "freehand" technique, but no prior study has assessed for superiority between these 2 techniques. Furthermore, to-date assessment of post-operative reconstruction has not been tested in detail as post-THA assessments are based on radiographs which provide incomplete, 2-dimensional, assessments and are lacking the important axial plane reconstruction parameters. The aims of this prospective, randomized, trial are to 1. appraise the ability to achieve the pre-operative 3-D plan (as per FormusLab) through a comparison of pre-op plan to post-operative reconstruction; 2. compare ability to accurately reconstruct hip following THA between "navigated-" (IntelliJoint®) and "measured-" techniques; and in doing so it will also 3. assess the accuracy of the intra-operative assessments of reconstruction through a comparison of objective (i.e. measured) intra-operative assessments with the post-operative reconstructions achieved.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are signed for a THA for primary or secondary osteoarthritis without overt deformity that would require revision type implants and with good enough bone quality to be listed for uncemented component implantation.

Exclusion Criteria:

* Secondary OA due to Dysplasia (Hartofilakidis >1)
* Avascular necrosis of the hip with destruction of joint structure
* Sequelae of Pediatric deformity with abnormal anatomy
* Cemented fixation of femur or acetabulum
* Previous arthroplasty-type procedure
* Previous septic arthritis of the hip

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Assessment - Oxford Hip Score | once pre-operatively and once one-year post-operatively
  The Oxford Hip Score will be given to patients to assess subjective measures of hip pain. Scores for each question from 0 to 4 with 4 being the best outcome. This method, when summed, produces overall scores running from 0 to 48 with 48 being the best outcome
Change in mobility, self-care, usual activities, pain/discomfort and anxiety/depression- EuroQol | once pre-operatively and once one-year post-operatively
  the EuroQol (EQ-5D-5L) will be given to patients to assess subjective measures mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems.
Change in physical, mental, and social health- PROMIS Global-10 | once pre-operatively and once one-year post-operatively
  the PROMIS Global-10 will be given to patients to assess subjective measures of physical, mental and social health. It is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. Higher scores indicate worse physical and mental health
Adverse Events | 90 days post-operatively
  Serious adverse events will be monitored. This includes:
  * Wound complication
  * Dislocation
  * Fracture
  * Infection
  * Re-operation
  * Revision surgery

SECONDARY OUTCOMES:
Accuracy of reconstruction (in mm) | post-operatively (within one week post-operatively)
  A measure (in mm) of how close the planned to actual reconstruction using the aforementioned reconstruction parameters. This will be assessed using:
  * Acetabular component orientation
  * Accuracy of acetabular component orientation
    o Accuracy of femoral version restoration
  * Combined version of arthroplasty in degrees
    * Accuracy of combined version restoration
  * Femoral Offset in mm
    o Accuracy of achieving femoral offset
  * Acetabular offset in mm
    o Accuracy of achieving acetabular offset
  * Total offset in mm
    o Accuracy of achieving total offset
  * Leg Length in mm o Accuracy of achieving leg length
Comparison of margin of error | Through study completion, an average of 1 year
  This outcome will measure what the margin of error is between intra-operatively measured values and those determined from the post-operative CT scan. This will be done using statistical analysis of data for patients in both study arms.
Accuracy of reconstruction on outcome | Through study completion, an average of 1 year
  This outcome measure will assess the accuracy of reconstruction correlate with outcome (adverse events and PROMs). This will be done by analyzing accuracy as depicted by the variables in outcome measure 5, and how these measures of accuracy correlate to patient reported outcome measure scores and rates of adverse events
Accuracy of reconstruction (in degrees) | post-operatively (within one week post-operatively)
  A measure (in degrees) of how close the planned to actual reconstruction using the aforementioned reconstruction parameters. This will be assessed using:
  Acetabular component orientation (Radiographic inclination/anteversion in degrees as per Murray)
  * Accuracy of acetabular component orientation (i.e. deviation from target - aim for deviation of < ±5˚)
    ● Femoral Component Version in degrees
  * Accuracy of femoral version restoration (aim for version difference to be less than ±5˚ from pre-operative plan)
    ● Combined version of arthroplasty in degrees
  * Accuracy of combined version restoration (sum of acetabular and femoral version; aim for combined version to be less than ±10˚ from pre-operative plan)

CONTACTS AND LOCATIONS:
Overall Officials: George Grammatopoulos, MD, Principal Investigator — The Ottawa Hospital

REFERENCES:
- [Background] Fang CJ, Shaker JM, Ward DM, Jawa A, Mattingly DA, Smith EL. Financial Burden of Revision Hip and Knee Arthroplasty at an Orthopedic Specialty Hospital: Higher Costs and Unequal Reimbursements. J Arthroplasty. 2021 Aug;36(8):2680-2684. doi: 10.1016/j.arth.2021.03.044. Epub 2021 Mar 23. PMID 33840537
- [Background] Hu X, Zheng N, Chen Y, Dai K, Dimitriou D, Li H, Tsai TY. Optimizing the Femoral Offset for Restoring Physiological Hip Muscle Function in Patients With Total Hip Arthroplasty. Front Bioeng Biotechnol. 2021 Mar 30;9:645019. doi: 10.3389/fbioe.2021.645019. eCollection 2021. PMID 33869155
- [Background] Grammatopoulos G, Thomas GE, Pandit H, Beard DJ, Gill HS, Murray DW. The effect of orientation of the acetabular component on outcome following total hip arthroplasty with small diameter hard-on-soft bearings. Bone Joint J. 2015 Feb;97-B(2):164-72. doi: 10.1302/0301-620X.97B2.34294. PMID 25628277
- [Background] Agarwal S, Eckhard L, Walter WL, Peng A, Hatton A, Donnelly B, de Steiger R. The Use of Computer Navigation in Total Hip Arthroplasty Is Associated with a Reduced Rate of Revision for Dislocation: A Study of 6,912 Navigated THA Procedures from the Australian Orthopaedic Association National Joint Replacement Registry. J Bone Joint Surg Am. 2021 Oct 20;103(20):1900-1905. doi: 10.2106/JBJS.20.00950. PMID 34143758
- [Background] Shon WY, Baldini T, Peterson MG, Wright TM, Salvati EA. Impingement in total hip arthroplasty a study of retrieved acetabular components. J Arthroplasty. 2005 Jun;20(4):427-35. doi: 10.1016/j.arth.2004.09.058. PMID 16124957
- [Background] Barrack RL, Krempec JA, Clohisy JC, McDonald DJ, Ricci WM, Ruh EL, Nunley RM. Accuracy of acetabular component position in hip arthroplasty. J Bone Joint Surg Am. 2013 Oct 2;95(19):1760-8. doi: 10.2106/JBJS.L.01704. PMID 24088968
- [Background] Callanan MC, Jarrett B, Bragdon CR, Zurakowski D, Rubash HE, Freiberg AA, Malchau H. The John Charnley Award: risk factors for cup malpositioning: quality improvement through a joint registry at a tertiary hospital. Clin Orthop Relat Res. 2011 Feb;469(2):319-29. doi: 10.1007/s11999-010-1487-1. PMID 20717858
- [Background] Bosker BH, Verheyen CC, Horstmann WG, Tulp NJ. Poor accuracy of freehand cup positioning during total hip arthroplasty. Arch Orthop Trauma Surg. 2007 Jul;127(5):375-9. doi: 10.1007/s00402-007-0294-y. Epub 2007 Feb 13. PMID 17297597
- [Background] Schwarzkopf R, Muir JM, Paprosky WG, Seymour S, Cross MB, Vigdorchik JM. Quantifying Pelvic Motion During Total Hip Arthroplasty Using a New Surgical Navigation Device. J Arthroplasty. 2017 Oct;32(10):3056-3060. doi: 10.1016/j.arth.2017.04.046. Epub 2017 May 4. PMID 28559196
- [Background] Pongkunakorn A, Chatmaitri S, Diewwattanawiwat K. Use of smartphone to improve acetabular component positioning in total hip athroplasty: A comparative clinical study. J Orthop Surg (Hong Kong). 2019 Jan-Apr;27(1):2309499019825578. doi: 10.1177/2309499019825578. PMID 30798733
- [Background] Gupta R, Pathak P, Singh R, Majumdar KP. Double-Stitch Technique: A Simple and Effective Method to Minimize Limb Length Discrepancy after Total Hip Arthroplasty. Indian J Orthop. 2019 Jan-Feb;53(1):169-173. doi: 10.4103/ortho.IJOrtho_188_18. PMID 30905998
- [Background] Mitsutake R, Tanino H, Nishida Y, Higa M, Ito H. A simple angle-measuring instrument for measuring cemented stem anteversion during total hip arthroplasty. BMC Musculoskelet Disord. 2020 Feb 19;21(1):113. doi: 10.1186/s12891-020-3142-7. PMID 32075628
- [Background] Steppacher SD, Kowal JH, Murphy SB. Improving cup positioning using a mechanical navigation instrument. Clin Orthop Relat Res. 2011 Feb;469(2):423-8. doi: 10.1007/s11999-010-1553-8. PMID 20852974
- [Background] Meermans G, Van Doorn WJ, Koenraadt K, Kats J. The use of the transverse acetabular ligament for determining the orientation of the components in total hip replacement: a randomised controlled trial. Bone Joint J. 2014 Mar;96-B(3):312-8. doi: 10.1302/0301-620X.96B3.32989. PMID 24589784
- [Background] Paprosky WG, Muir JM. Intellijoint HIP(R): a 3D mini-optical navigation tool for improving intraoperative accuracy during total hip arthroplasty. Med Devices (Auckl). 2016 Nov 18;9:401-408. doi: 10.2147/MDER.S119161. eCollection 2016. PMID 27920583
- [Background] Parvizi J, Benson JR, Muir JM. A new mini-navigation tool allows accurate component placement during anterior total hip arthroplasty. Med Devices (Auckl). 2018 Mar 22;11:95-104. doi: 10.2147/MDER.S151835. eCollection 2018. PMID 29606894
- [Background] Kievit AJ, Dobbe JGG, Mallee WH, Blankevoort L, Streekstra GJ, Schafroth MU. Accuracy of cup placement in total hip arthroplasty by means of a mechanical positioning device: a comprehensive cadaveric 3d analysis of 16 specimens. Hip Int. 2021 Jan;31(1):58-65. doi: 10.1177/1120700019874822. Epub 2019 Sep 11. PMID 31506002
- [Background] Snijders T, van Gaalen SM, de Gast A. Precision and accuracy of imageless navigation versus freehand implantation of total hip arthroplasty: A systematic review and meta-analysis. Int J Med Robot. 2017 Dec;13(4). doi: 10.1002/rcs.1843. Epub 2017 May 29. PMID 28556582
- [Background] Singh V, Realyvasquez J, Simcox T, Rozell JC, Schwarzkopf R, Davidovitch RI. Robotics Versus Navigation Versus Conventional Total Hip Arthroplasty: Does the Use of Technology Yield Superior Outcomes? J Arthroplasty. 2021 Aug;36(8):2801-2807. doi: 10.1016/j.arth.2021.02.074. Epub 2021 Mar 5. PMID 33773864
- [Background] Koper MC, Reijman M, van Es EM, Waarsing JH, Koot HWJ, Keizer SB, Jansen I, van Biezen FC, Verhaar JAN, Bos PK. No added value for Computer-Assisted surgery to improve femoral component positioning and Patient Reported Outcomes in Hip Resurfacing Arthroplasty; a multi-center randomized controlled trial. BMC Musculoskelet Disord. 2019 Oct 25;20(1):473. doi: 10.1186/s12891-019-2883-7. PMID 31651318
- [Background] Innmann MM, Maier MW, Streit MR, Grammatopoulos G, Bruckner T, Gotterbarm T, Merle C. Additive Influence of Hip Offset and Leg Length Reconstruction on Postoperative Improvement in Clinical Outcome After Total Hip Arthroplasty. J Arthroplasty. 2018 Jan;33(1):156-161. doi: 10.1016/j.arth.2017.08.007. Epub 2017 Aug 12. PMID 28887022
- [Background] Schiffner E, Latz D, Jungbluth P, Grassmann JP, Tanner S, Karbowski A, Windolf J, Schneppendahl J. Is computerised 3D templating more accurate than 2D templating to predict size of components in primary total hip arthroplasty? Hip Int. 2019 May;29(3):270-275. doi: 10.1177/1120700018776311. Epub 2018 May 20. PMID 29781288
- [Background] Minoda Y, Ohzono K, Aihara M, Umeda N, Tomita M, Hayakawa K. Are acetabular component alignment guides for total hip arthroplasty accurate? J Arthroplasty. 2010 Sep;25(6):986-9. doi: 10.1016/j.arth.2009.07.016. Epub 2009 Oct 17. PMID 19837559
- [Background] Beverland DE, O'Neill CK, Rutherford M, Molloy D, Hill JC. Placement of the acetabular component. Bone Joint J. 2016 Jan;98-B(1 Suppl A):37-43. doi: 10.1302/0301-620X.98B1.36343. PMID 26733639
- [Background] Bonnin MP, Archbold PH, Basiglini L, Fessy MH, Beverland DE. Do we medialise the hip centre of rotation in total hip arthroplasty? Influence of acetabular offset and surgical technique. Hip Int. 2012 Jul-Aug;22(4):371-8. doi: 10.5301/HIP.2012.9350. PMID 22865253
- [Background] Merle C, Innmann MM, Waldstein W, Pegg EC, Aldinger PR, Gill HS, Murray DW, Grammatopoulos G. High Variability of Acetabular Offset in Primary Hip Osteoarthritis Influences Acetabular Reaming-A Computed Tomography-Based Anatomic Study. J Arthroplasty. 2019 Aug;34(8):1808-1814. doi: 10.1016/j.arth.2019.03.065. Epub 2019 Apr 1. PMID 31122846
- [Background] Meermans G, Goetheer-Smits I, Lim RF, Van Doorn WJ, Kats J. The difference between the radiographic and the operative angle of inclination of the acetabular component in total hip arthroplasty: use of a digital protractor and the circumference of the hip to improve orientation. Bone Joint J. 2015 May;97-B(5):603-10. doi: 10.1302/0301-620X.97B5.34781. PMID 25922452
- [Background] Lee YK, Kim JW, Kim TY, Ha YC, Koo KH. Validity of the intra-operative measurement of stem anteversion and factors for the erroneous estimation in cementless total hip arthroplasty using postero-lateral approach. Orthop Traumatol Surg Res. 2018 May;104(3):341-346. doi: 10.1016/j.otsr.2017.11.023. Epub 2018 Feb 16. PMID 29458202
- [Background] Dorr LD, Wan Z, Malik A, Zhu J, Dastane M, Deshmane P. A comparison of surgeon estimation and computed tomographic measurement of femoral component anteversion in cementless total hip arthroplasty. J Bone Joint Surg Am. 2009 Nov;91(11):2598-604. doi: 10.2106/JBJS.H.01225. PMID 19884433
- [Background] Blumenfeld TJ. Pearls: Clinical Application of Ranawat's Sign. Clin Orthop Relat Res. 2017 Jul;475(7):1789-1790. doi: 10.1007/s11999-017-5376-8. Epub 2017 May 11. No abstract available. PMID 28497375
- [Background] Dorr LD, Malik A, Dastane M, Wan Z. Combined anteversion technique for total hip arthroplasty. Clin Orthop Relat Res. 2009 Jan;467(1):119-27. doi: 10.1007/s11999-008-0598-4. Epub 2008 Nov 1. PMID 18979146
- [Background] Amuwa C, Dorr LD. The combined anteversion technique for acetabular component anteversion. J Arthroplasty. 2008 Oct;23(7):1068-70. doi: 10.1016/j.arth.2008.04.025. Epub 2008 Jun 4. PMID 18534533
- [Background] Ogawa T, Takao M, Hamada H, Sakai T, Sugano N. Soft tissue tension is four times lower in the unstable primary total hip arthroplasty. Int Orthop. 2018 Sep;42(9):2059-2065. doi: 10.1007/s00264-018-3908-9. Epub 2018 Mar 27. PMID 29589084
- [Background] Hill JC, Archbold HA, Diamond OJ, Orr JF, Jaramaz B, Beverland DE. Using a calliper to restore the centre of the femoral head during total hip replacement. J Bone Joint Surg Br. 2012 Nov;94(11):1468-74. doi: 10.1302/0301-620X.94B11.29144. PMID 23109624
- [Background] Dorr LD, Hishiki Y, Wan Z, Newton D, Yun A. Development of imageless computer navigation for acetabular component position in total hip replacement. Iowa Orthop J. 2005;25:1-9. PMID 16089064
- [Background] Jacob I, Benson J, Shanaghan K, Gonzalez Della Valle A. Acetabular positioning is more consistent with the use of a novel miniature computer-assisted device. Int Orthop. 2020 Mar;44(3):429-435. doi: 10.1007/s00264-020-04484-2. Epub 2020 Jan 22. PMID 31965312
- [Background] Christ A, Ponzio D, Pitta M, Carroll K, Muir JM, Sculco PK. Minimal Increase in Total Hip Arthroplasty Surgical Procedural Time with the Use of a Novel Surgical Navigation Tool. Open Orthop J. 2018 Sep 28;12:389-395. doi: 10.2174/1874325001812010389. eCollection 2018. PMID 30416609
- [Background] Murray DW. The definition and measurement of acetabular orientation. J Bone Joint Surg Br. 1993 Mar;75(2):228-32. doi: 10.1302/0301-620X.75B2.8444942.
- [Background] Gross AE, Safir OA, Kuzyk PRT, Sculco PK, Wolfstadt J, Girardi BL, et al. Optimizing leg length and cup position: A surgical navigation tool. Seminars in Arthroplasty. 2018;29(3):157-60.